CLINICAL TRIAL: NCT01627795
Title: A Single-center, Open Label Study for Evaluation of the Safety and Efficacy of Oshadi D and Oshadi R for Malignant Mesothelioma Treatment - A Phase IIa Study
Brief Title: Safety and Efficacy of Oshadi D and Oshadi R for Malignant Mesothelioma Treatment
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oshadi Drug Administration (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OS-MES-P2-01
Record Dates: First submitted 2012-06-20; First posted 2012-06-26 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Mesothelioma
Keywords: Malignant Mesothelioma; Cancer; Anti cancer agents
MeSH Terms: conditions — Mesothelioma; Mesothelioma, Malignant; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oshadi D and Oshadi R (Experimental): anti cancer agents
  Interventions: Drug: Oshadi D and Oshadi R

INTERVENTIONS:
Drug: Oshadi D and Oshadi R — anti cancer agents

SUMMARY:
Malignant mesothelioma is a rare neoplasm that arises most commonly from the mesothelial surfaces of the pleural cavity, occasionally from the peritoneal surface, and rarely from the tunica vaginalis or pericardium. It has an extremely poor prognosis with a median survival of 4 to 13 months for untreated patients 1 and 6 to 18 months for treated patients, regardless of the therapeutic approach.

The anticancer activity of Oshadi D and Oshadi R treatment was tested in preclinical studies and in phase I clinical study. Four metastatic mesothelioma patients are treated for 5 to 12 months. The Oshadi D and Oshadi R combination treatment was generally well-tolerated with no dose-limiting toxicities observed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven diagnosis of malignant mesothelioma
* Man or woman 21 years and above
* Adequate performance status (ECOG 0, 1, or 2)
* Patient must have adequate organ function as the following:

  * Absolute neutrophils counts (ANS) > 2500/μL.
  * Platelets > 150,000/μL.
  * Hemoglobin > 10 g/dL.
  * Total Bilirubin < 1.5 Upper Normal Limit (UNL).
  * Alanine aminotransferase (ALT), AST (aspartate aminotransferase)and alkaline phosphatase must be < 1.5 times of the upper limit of normal.
  * LDH (lactate dehydrogenase) < 500 int. unit/L
  * Estimated GFR (glomerular filtration rate) > 45 ml/min.
* Written informed consent
* Females of childbearing potential and males must be willing to use an effective method of contraception (hormonal or barrier method of birth control; abstinence) from the time consent is signed until 6 weeks after treatment discontinuation.
* Females of childbearing potential must have a negative pregnancy test within 7 days prior to being registered for protocol therapy.

Exclusion Criteria:

* Evidence of liver metastasis
* Any bone involvement
* Prior radiotherapy, cytotoxic or biologic systemic treatment
* Any history of Asthma or COPD (chronic obstructive pulmonary disease) that needs systemic therapy with steroids for more than 2 weeks during the last 2 years.
* Treatment with systemic steroids for more then 1 month during the last year.
* Active smokers that are unable to quite smoking
* Any treatment with investigational agent within 30 days prior to registration for protocol therapy.
* Cerebrovascular accident, transient ischemic attack or myocardial infarction within 6 months prior to registration for protocol therapy.
* Evidence of pulmonary embolism within 6 months prior to registration for protocol therapy.
* Any history of solid or hematologic malignancies.
* Patient with positive HIV serology at screening.
* Female patient who are breastfeeding or have a positive pregnancy test at screening or at any time during the study.
* Uncontrolled hypertension (> 150/100 mm Hg despite optimal medical therapy).
* Evidence of ongoing cardiac dysrhythmias of NCI CTCAE (Common Toxicity Criteria for Adverse Effects) Version 3.0 grade 2.
* Patients in whom radiation or surgery is indicated
* Significant swallowing disorders.
* Small bowel surgery.
* Suspicion of absorption disruption as a result of abdominal radiation
* Pre-existing malabsorption syndrome, irritable bowel syndrome or other clinical situation which could affect oral absorption.
* Evidence of concurrent (< 5 years) second malignancy
* Mental disorders.
* Inability to give written informed consent.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-08 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events and serious adverse events occurence | One month following treatment initiation
  Adverse events and serious adverse events report

SECONDARY OUTCOMES:
overall survival time | 12 months
  Overall survival time from treatment initiation

CONTACTS AND LOCATIONS:
Overall Officials: Hovav Nehushtan, Prof., Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel